CLINICAL TRIAL: NCT00299923
Title: Randomized, Open-Label, Multicenter Study Examining the Effects of Duration of Treatment of PEGASYS® in Combination With Daily COPEGUS® + Amantadine in Patients With Chronic HCV After Relapse to Previous (Peg)IFN + Ribavirin Therapy.
Brief Title: Study for Patients With Chronic HCV (GT 1 or 3) Who Relapsed to Previous (Peg)Interferon/ Ribavirin Combination Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Hamburg-Eppendorf (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Hoffmann-La Roche (Industry)
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML 18545 (TRELA); EudraCT-Nr.: 2005-001207-19
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: Hepatitis C, Chronic; Relapse
Keywords: drug therapy; Interferon
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence | interventions — peginterferon alfa-2a; Ribavirin; Amantadine

INTERVENTIONS:
Drug: Peginterferon alfa-2a, Ribavirin, Amantadine

SUMMARY:
The aim of this study is, to compare the relapse rate in chronic HCV patients with genotype 1 or 3 under the combination of standard dose Peg-Interferon alfa-2a (PEG-IFN alfa-2a), Ribavirin (RBV) and Amantadine (AMA) given for 72 weeks (group A), versus the same combination, given for 48 weeks (group B) in patients who relapsed to previous combination therapy to conventional or pegylated (PEG) Interferon alfa and Ribavirin. Relapse ist defined as percentage of patients with non-detectable HCV-RNA at end of therapy (week 48 GT1/ week 24 GT 3) who become HCV-RNA positive during a follow-up period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Relapsers to previous combination therapy with (PEG-)IFN alfa-/Ribavirin and a negative HCV-RNA test result at the end of this regular treatment course and positive HCV-RNA test result during the follow-up period.
* Termination of (PEG-)IFN alfa-/ribavirin therapy at least 3 months prior to enrolment
* Chronic HCV infection genotype 1 or 3.
* Serum HCV-RNA quantifiable at >100 IU/mL by COBAS AmpliPrep or another quantitative HCV-RNA PCR test (reported in IU)
* Compensated liver disease (Child-Pugh A)
* Exclusion of HCC in patients with cirrhosis or transition to cirrhosis. In patients with AFP >50 ng/mL an established assay for exclusion of HCC has to be done
* Negative urine or blood pregnancy test
* All fertile males and females must use two reliable forms of effective contraception (combined) during treatment with study drugs and 6 months post treatment

Exclusion Criteria (at screening):

* Hypersensitiveness to Interferon, PEG-IFN alfa-2a, Ribavirin and Amantadine or other ingredient of the drugs
* Ongoing pregnancy or breast feeding
* Male partners of women who are pregnant or with women without effective contraception
* Signs or symptoms of hepatocellular carcinoma
* Chronic HCV infection genotype 2, 4, 5 or 6
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment < 6 months prior to the first dose of study drug and during study period. Exception: patients who have had a limited (< 7 days) course of acyclovir or valacyclovir for herpetic lesions < 1 month prior to the first administration of test drug are not excluded.
* Any investigational drug < 6 weeks prior to the first dose of study drug
* Positive test for anti-HAV IgM, HBsAg, anti-HBc IgM, anti-HIV
* History or other evidence of a medical condition associated with chronic liver disease other than HCV
* History or other evidence of decompensated liver disease or a Child-Pugh score > 6.
* Hb <12 g/dL (<120 g/L) in women or <13 g/dL (<130 g/L) in men at screening
* Any patient with an increased baseline risk for anemia or for whom anemia would be medically problematic
* Neutrophil count <1,500 cells/mm3 and/or platelet count <90,000 cells/mm3
* Serum creatinin concentration >1.5 mg/dl
* History of severe psychiatric disease, especially depression.
* History of a severe seizure disorder that can not be stabilized by medication
* History of immunologically mediated disease
* Chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease
* History of major organ transplantation except corneatransplantation
* Evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Thyroid dysfunction not adequately controlled
* Evidence of severe retinopathy or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Evidence of active drug abuse within one year of study entry except of a prescribed stable opioid substitution
* Take of Memantine during study period
* Cardiomyopathy and myocarditis
* AV-Block II° and III°
* Pre-existing bradycardia < 55 counts/min
* Known QT-interval (QTc after Bazett > 420 ms) or recognized U-waves or congenital QT-syndrome
* History of severe ventricular arrhythmia incl. Torsade de pointes
* Simultaneous therapy with Budipin or other medicine that extend the QT-interval like (e.g.antiarrhythmic drugs class IA and class III, antipsychotic drugs, tri- and tetracyclic antidepressants, antihistaminics, macrolide, gyrase inhibitors, Azol-antimykotics)
* Patients with obstructive glaucoma
* Patients with excitableness and confusion
* Patients with delirium and exogenic psychosis in the anamnesis
* Prostataadenome
* Diuretic medication of the type combination Triamterene/ Hydrochlorothiazide
* Inability or unwillingness to provide informed consent or abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-11

PRIMARY OUTCOMES:
- Comparison of the rate of relapse under the combination of standard dose PegIFN alfa-2a, Ribavirin and Amantadine given for 72 vs. 48 weeks.

SECONDARY OUTCOMES:
relationship between EVR during the first twelve weeks and SVR
virological response to the combination of standard dose defined as reduction of HCV RNA at week 4, 12, 24, 48 and 72 of treatment, separated between HCV-Genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Buggisch, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Medizinische Klinik 1
Locations (27):
- Germany (27):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Mannheim, Baden-Würtemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Württembeg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum rechts der Isar der TU München, München, Bavaria
  - Krankenhaus Barmherzige Brüder, Regensburg, Bavaria
  - Klinikum der Universität Regensburg, Regensburg, Bavaria
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Klinikum Bremen-Mitte, Bremen, City state Bremen
  - J. W.-Goethe-Universität, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universität Rostock, Rostock, Mecklenburg-Vorpommern
  - Klinikum der Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Klinikum der Universität Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinkum Münster, Münster, North Rhine-Westphalia
  - St-Josef-Hospital, Oberhausen, North Rhine-Westphalia
  - Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Bad Homburg/ Saar, Saarland
  - Klinikum der Medizinischen Fakultät der Martin-Luther Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Praxis Möller/ Heyne, Berlin, State of Berlin
  - Charité, Campus Benjamin Franklin, Berlin, State of Berlin
  - Charité, Campus Virchow-Klinikum, Med. Klinik (Gastroenterologie/ Hepatologie), Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Med. Klinik 1, Hamburg